CLINICAL TRIAL: NCT05965362
Title: Prognosis of Patients With Infective Endocarditis and Risk Stratification Value of Biomarkers (ENDEAVOR): a National Multi-center, Retrospective-prospective, Cohort Study Initiated by the Investigators
Brief Title: Prognosis of Patients With Infective Endocarditis and Risk Stratification Value of Biomarkers (ENDEAVOR）
Acronym: ENDEAVOR
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 521 Hospital of NORINCO Group (Other); Shaanxi Provincial People's Hospital (Other); Xiangyang Central Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-151
Record Dates: First submitted 2023-02-14; First posted 2023-07-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Infective Endocarditis
Keywords: Infective Endocarditis; Prognosis; Major Adverse Cardiac and Cerebrovascular event
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, feces, urine, valvular, superfluous organisms, adipose tissue and pericardial effusion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infective endocarditis group: Patients diagnosed with infective endocarditis.
  Interventions: Other: Observational; No Interventions were given.

INTERVENTIONS:
Other: Observational; No Interventions were given. — Observational; No Interventions were given.

SUMMARY:
In this study, by establishing a clinical cohort of infective endocarditis, we observed the natural prognosis and influencing factors in the process of disease development and regression; we used multi-omics technology to understand the prognostic value of its biomarkers, and provided new ideas and evidence for the pathogenesis, clinical diagnosis and treatment of IE.

DETAILED DESCRIPTION:
Infective endocarditis is an inflammation of the inner lining of the heart valves or ventricular walls caused by direct infection of the heart by bacteria, fungi and other microorganisms via the bloodstream route. At present, the clinical diagnosis of IE is mainly based on a combination of typical symptoms, imaging and blood culture, etc. Finding more sensitive means and more accurate indicators for early detection of IE flora distribution characteristics is of great significance for the prevention and targeted treatment of IE. Therefore, in this study, by establishing a clinical cohort of infective endocarditis, we observed the natural prognosis and influencing factors in the process of disease development and regression; we used multi-omics technology to understand the prognostic value of its biomarkers, and provided new ideas and evidence for the pathogenesis, clinical diagnosis and treatment of IE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically confirmed infective endocarditis

Exclusion Criteria:

* Patients refuse to sign informed consent form
* Patients who combined with serious systemic diseases, cannot tolerate the acquisition of biological samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically confirmed infective endocarditis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of MACCE | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  MACCE is major adverse cardio-cerebrovascular events, including myocardial infarction, stroke, vessel revascularization and all-cause death. The MACCE will be assessed from the medical records.

SECONDARY OUTCOMES:
Incidence of adverse thrombus complications | 5 years after the enrollment.
  Adverse thrombus complications including systemic embolism, infected aneurysm, splenic abscess, etc.
Change in the incidence of infection recurrence | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  Diagnosis of infective endocarditis by clinical guidelines, which will be assessed from medical records.
Change in the incidence of myocardial infarction | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  Myocardial infarction, diagnosed by clinical doctors, will be assessed from medical records.
Change in the incidence of stroke | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  Stroke, diagnosed by clinical doctors, will be assessed from medical records.
Change in the incidence of vessel revascularization | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  Vessel revascularization, diagnosed by clinical doctors, will be assessed from medical records.
Change in the incidence of all-cause death | 1, 3, 6 months and 1, 2, 3, 5 years after enrollment.
  All-cause death, diagnosed by clinical doctors, will be assessed from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China